CLINICAL TRIAL: NCT03123614
Title: Efficacy and Safety of Loteprednol 0.5% Gel for Routine Prophylaxis After Photorefractive Keratectomy Compared to Prednisolone Acetate 1% Suspension and Fluorometholone 0.1% Suspension
Brief Title: Loteprednol vs. Prednisolone and Fluorometholone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Mark Mifflin, Professor, Ophthalmology/Visual Sciences, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 75978
Record Dates: First submitted 2017-04-17; First posted 2017-04-21 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Intraocular Pressure; Corneal Opacity
Keywords: Photorefractive keratectomy
MeSH Terms: conditions — Corneal Opacity | interventions — Loteprednol Etabonate; prednisolone acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Examiners are masked to the treatment arm when obtaining measurements of intraocular pressure (IOP) and grading corneal haze.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Loteprednol Etabonate 0.5% Oph Gel (Active Comparator): Group 1 will use loteprednol 0.5% gel in both eyes, starting at a frequency of four times per day for the first week and then tapered off based on clinical judgement of the corneal healing response.
  Interventions: Drug: Loteprednol Etabonate 0.5% Oph Gel
- Prednisolone acetate 1% Oph Susp (Active Comparator): Group 2 will use prednisolone acetate 1% suspension in both eyes, starting at a frequency of four times per day for the first week, then tapered down to a regimen of fluorometholone 0.1% suspension, which will then be tapered off based on clinical judgement of the corneal healing response.
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp

INTERVENTIONS:
Drug: Loteprednol Etabonate 0.5% Oph Gel
  Arms: Loteprednol Etabonate 0.5% Oph Gel
Drug: Prednisolone Acetate 1% Oph Susp
  Arms: Prednisolone acetate 1% Oph Susp

SUMMARY:
Corneal haze, in which the cornea becomes cloudy, is a well-known and a potentially vision-threatening postoperative complication of photorefractive keratectomy (PRK). Topical ophthalmic corticosteroids are routinely prescribed by most surgeons postoperatively to help prevent this complication.

Goals of topical steroids use after PRK include effective modulation of the healing response to prevent corneal haze while at the same time minimizing side effects, such as intraocular pressure elevation or cataract formation. Loteprednol etabonate is a corticosteroid that exerts its therapeutic effects and is then quickly changed into inactive metabolites. This relatively fast metabolism of loteprednol gives it a lower side effect profile than other steroids, including a smaller effect on intraocular pressure. In the ophthalmic literature, there is currently no consensus on a standard regimen or which type of corticosteroid should be used after PRK.

Investigators are conducting a prospective, randomized trial to compare the incidence of intraocular pressure rise and visually significant postoperative corneal haze after PRK with the use of loteprednol 0.5% gel compared to the use of earlier generation steroids, prednisolone acetate 1% suspension and fluorometholone 0.1% suspension.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who are deemed suitable candidates for PRK after routine refractive surgery screening will be considered eligible for participation in this study.
* Subjects must be at least 21 years of age and not pregnant or nursing (due to fluctuations in visual parameters during pregnancy).

Exclusion Criteria:

* Selection will be consistent with the current standard of care for PRK. Any patient that is not a suitable candidate for PRK will not be included.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mifflin, MD, Principal Investigator — University of Utah Moran Eye Center
Locations (1):
- Moran Eye Center - Midvalley Location, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Loteprednol Etabonate 0.5% Oph Gel: Group 1 will use loteprednol 0.5% gel in both eyes, starting at a frequency of four times per day for the first week and then tapered off based on clinical judgement of the corneal healing response.
  Loteprednol Etabonate 0.5% Oph Gel
- Prednisolone Acetate 1% Oph Susp: Group 2 will use prednisolone acetate 1% suspension in both eyes, starting at a frequency of four times per day for the first week, then tapered down to a regimen of fluorometholone 0.1% suspension, which will then be tapered off based on clinical judgement of the corneal healing response.
  Prednisolone Acetate 1% Oph Susp
Period: Overall Study
Arm/Group | Loteprednol Etabonate 0.5% Oph Gel | Prednisolone Acetate 1% Oph Susp
Started | 57; 114 Eyes | 74; 147 Eyes
Completed | 57; 114 Eyes | 74; 147 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol Etabonate 0.5% Oph Gel | Prednisolone Acetate 1% Oph Susp | Total
Number analyzed (Participants) | 57 | 74 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 74 | 131
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (8.8) | 35.3 (6.2) | 35.0 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 36 | 60
  Male | 33 | 38 | 71
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 74 | 131
Intraocular Pressure [Mean (Standard Deviation); unit: mmHg] | 14.38 (2.11) | 14.30 (2.13) | 14.34 (2.12)

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP) From Baseline Through Month 3
Description: Intraocular pressure will be measured by applanation tonometry
Time Frame: Baseline, 1 week post-op, 1 month post-op, 2 months post-op, 3 months post-op
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Loteprednol Etabonate 0.5% Oph Gel | Prednisolone Acetate 1% Oph Susp
Number analyzed (Participants) | 57 | 74
mmHg
  Baseline intraocular pressure (IOP) | 14.38 (2.11) | 14.30 (2.13)
  IOP 1 week postop | 13.67 (2.34) | 13.28 (3.37)
  IOP 1 month postop | 14.15 (2.88) | 14.60 (4.20)
  IOP 2 months postop | 13.36 (2.53) | 13.16 (2.80)
  IOP 3 months postop | 13.15 (2.43) | 12.22 (2.38)

2. Secondary Outcome: Number of Eyes With Corneal Haze
Description: As determined by slit lamp examination
Time Frame: 12 months
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Loteprednol Etabonate 0.5% Oph Gel | Prednisolone Acetate 1% Oph Susp
Number analyzed (Participants) | 57 | 74
Number analyzed (Eyes) | 114 | 147
Eyes | 3 | 7

3. Secondary Outcome: Uncorrected Visual Acuity
Description: Best uncorrected visual acuity will be measured at 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Loteprednol Etabonate 0.5% Oph Gel | Prednisolone Acetate 1% Oph Susp
Number analyzed (Participants) | 57 | 74
logMAR | -0.078 (0.10) | -0.075 (0.09)

4. Secondary Outcome: Best Corrected Visual Acuity at 3 Months
Description: Best uncorrected visual acuity will be measured at 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Loteprednol Etabonate 0.5% Oph Gel | Prednisolone Acetate 1% Oph Susp
Number analyzed (Participants) | 57 | 74
logMAR | -0.120 (0.059) | -0.114 (0.03)

ADVERSE EVENTS:
Time Frame: 3 years and 10 months
Arm/Group | Loteprednol Etabonate 0.5% Oph Gel | Prednisolone Acetate 1% Oph Susp
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/74
Other Adverse Events (participants affected / at risk) | 3/57 | 7/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate 0.5% Oph Gel (N=57) | Prednisolone Acetate 1% Oph Susp (N=74)
Non-visually significant corneal haze (Eye disorders) | 3 (3) | 7 (7) — Cornea haze

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/14/NCT03123614/Prot_SAP_000.pdf